CLINICAL TRIAL: NCT02741713
Title: Analgesic Benefit of PECS Blocks for Biceps Tenodesis Shoulder Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00030173
Record Dates: First submitted 2016-04-07; First posted 2016-04-18 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Biceps Tendonitis
MeSH Terms: interventions — Solutions; Injections; Bupivacaine; Epinephrine; Clonidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interscalene Block plus Sham Block (Sham Comparator): Twenty subjects will receive an ultrasound guided interscalene nerve block using the Solution for Injection in Interscalene Block dosed at the upper trunk location near the 6th cervical vertebral level, per standard clinical practice. A Sham Block of in area of PECS "Pectoralis" block will be done to allow for assessment of the intervention. Using the Solution for Injection in Sham Block.
  Interventions: Procedure: Interscalene Block; Procedure: Sham Block; Drug: Solution for Injection in Interscalene Block; Drug: Solution for Injection in Sham Block
- Interscalene plus PECS Blocks (Active Comparator): Twenty patients will receive an ultrasound guided interscalene nerve block Solution for Injection in Interscalene Block dosed at the upper trunk location near the 6th cervical vertebral level, per standard clinical practice. For the Intervention, these subjects will also a PECS "Pectoralis" 1 and 2 Blocks using the Solution for Injection PECS Blocks, dosed at the PECS1 location and PECS2 location as described by Blanco, et al.
  Interventions: Procedure: PECS "Pectoralis" 1 and 2 Blocks; Procedure: Interscalene Block; Drug: Solution for Injection in Interscalene Block; Drug: Solution for Injection PECS Blocks

INTERVENTIONS:
Procedure: PECS "Pectoralis" 1 and 2 Blocks — An interscalene and a PECS "Pectoralis" 1 and 2 block will be performed on the subjects.
  Arms: Interscalene plus PECS Blocks
Procedure: Interscalene Block — An interscalene block will be performed on the subjects.
Procedure: Sham Block
  Arms: Interscalene Block plus Sham Block
Drug: Solution for Injection in Interscalene Block — 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine
  Other Names: bupivacaine; epinephrine; clonidine
Drug: Solution for Injection in Sham Block — Lidocaine 1%
  Other Names: Lidocaine
  Arms: Interscalene Block plus Sham Block
Drug: Solution for Injection PECS Blocks — 10mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at the PECS1 location and 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at the PECS2 location
  Other Names: bupivacaine; epinephrine; clonidine
  Arms: Interscalene plus PECS Blocks

SUMMARY:
The standard practice for arthroscopic shoulder surgery at our institution is a general anesthetic with a long-acting interscalene block for post-operative pain control, which can reduce the amount of opiates needed after surgery. The interscalene block is effective in providing analgesia to the majority of the shoulder joint and has been shown to reduce post-operative pain scores after arthroscopic shoulder surgeries. However, there is a subset of arthroscopic shoulder surgery patients who have pain in the axilla even in the setting of a functioning interscalene brachial plexus nerve block. One of our surgeons has reported a high incidence of axillary pain in patients who undergo a sub-pectoral biceps tenodesis as part of their arthroscopic procedure. A newly described nerve block approach to the nerves that supply sensation to the axillary region called the PECS "Pectoralis" 1 & 2 block may provide additional analgesia to these patients.

The purpose of this prospective, randomized, observer and patient blinded, single-center, sham block trial is to determine if the addition of PECS blocks to an interscalene block will reduce the severity of axillary pain following arthroscopic shoulder surgery that involves a sub-pectoral biceps tenodesis. Secondarily, the study will assess the duration of PECS 1 & 2 and whether the block reduces post-operative opioid usage. We hypothesize that the addition of the PECS 1 & 2 block will reduce the severity of axillary pain at 6hrs and reduce postoperative narcotic usage for the first 24 hours.

DETAILED DESCRIPTION:
Subjects that meet the inclusion criteria will be assigned a group by using a random numbers generator. All subjects will receive the standard practice at our institution of an interscalene brachial plexus block along with a general anesthetic. The intervention arm will get an additional local anesthetic block targeting nerves that we presume cover the axillary region (PECS "Pectoralis" 1 & 2). These nerves in the upper chest are the lateral branches of the 2nd to 5th intercostal nerves, which includes the intercostobrachial nerve. The anesthesiologist placing the nerve blocks will be un-blinded to perform the procedures. Both the surgeon and the Acute Pain Service anesthesiologist will be blinded as to whether or not the intervention was provided to any given subject. The Acute Pain Service team will remain blinded and collect the data outcomes.

Initially, pilot data was collected in a total of ten patients with five patients randomized to each arm. Primary endpoint was NRS "Numerical Rating Scale" of 0-10 at 6hrs after block placement. Our pilot data indicate that the mean NRS is about 5 for the control group, with a standard deviation of 1.4. Using a two-sided two-sample t test (an alpha of 0.05 and power of 0.95), we conservatively estimate that 14 subjects per arm will be needed to detect a clinically meaningful difference of 2 in NRS between the arms. We decided to plan enrollment of 20 subjects per arm for potential loss during this randomized, double-blinded, single-center, sham block trial.

* Potential subjects undergoing arthroscopy will have their electronic medical record reviewed by the study team to look for exclusion criteria. If the subject is excluded, then they will be added to the Screening Log with date and reason for their exclusion. If all inclusion criteria are met, then the subject will be approached in the Regional Anesthesia area for their consent. A copy of the consent will be given to the study subject. The other informed consent document will be maintained by the study team in the research files.
* Patients will be asked to provide baseline pain scores both, at rest and with movement, on a scale of 0-10 (0 being no pain and 10 being the worst pain). Preoperative opioid use including drug(s), dosage and frequency will be recorded. Randomization of patients will then occur through the use of sequentially numbered envelopes with only those directly involved in the care of the patient during block placement being aware of which arm of the study the patient has been randomized. Those members of the study team who will be collecting post-operative data will be blinded to the randomization.

Standard American Society of Anesthesiology monitors and oxygen will be applied. Unless there is a contraindication, each patient will receive 650mg "milligrams" of oral acetaminophen. To standardize the effect on postoperative pain, ketamine will not be given as a preoperative sedation medication or intraoperative medication. No long acting opioids will be given in the operating room or post-anesthesia care unit. Intraoperative fentanyl will be limited to 5 micrograms per kg "kilogram". Intraoperative dexamethasone will not be given for post-operative nausea/vomiting prophylaxis.

Subjects will be sedated as per usual practice and will also be blinded to their randomization. All peripheral nerve blocks will be performed by a resident or fellow under supervision by an attending anesthesiologist. The attending anesthesiologist may perform the procedures alone. All volumes and concentrations of nerve block mixtures administered will be identical to assist in the blinding process.

All 40 subjects will receive an ultrasound guided interscalene nerve block using 20mL "milliliters" of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at the upper trunk location near the 6th cervical vertebral level, per standard clinical practice. The intervention arm, consisting of 20 patients, will additionally receive the following: 10mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine at the PECS1 location and 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine at the PECS2 location as described by Blanco, et al.3,4 All procedures will be performed under a sterile technique including the use of chlorhexidine prep of the skin, sterile gloves, sterile ultrasound probe covers with sterile ultrasound gel, a cap and a mask. For the interscalene block, a 21 gauge 90mm "millimeter" stimulating block needle will be directed, under real-time ultrasound guidance, into the interscalene muscle space at the level of the 5th and 6th cervical nerve roots. Twenty mL of the above local anesthetic mixture will be dosed incrementally, aspirating every 5 mL, to surround the upper trunk of the brachial plexus. For the PECS 1 & 2 block, a 21 gauge 90mm stimulating block needle will be placed under real-time ultrasound guidance at approximately the level of the 4th and 5th ribs near the mid-axillary line. The needle will be advanced into a tissue plane between the serratus anterior muscle and the pectoralis minor muscle. Twenty mL of the same local anesthetic mixture will be dosed incrementally, every 5 mL, to spread within this PEC2 space. The needle will be withdrawn, following the first injection, to a tissue plane between the pectoralis minor and pectoralis major muscles. Ten mL of the same local anesthetic mixture will be dosed incrementally, every 5 mL, to spread within this PEC1 space.

Fifteen and 30 minutes (if no change at 15min) following block placement, success will be assessed by absence/decrease of pin-prick sensation to a 25 gauge Whitacre needle in the following manner:

Cutaneous sensation will be tested over the deltoid region to assess for successful interscalene block.

Cutaneous sensation will be tested over the lateral aspect of the pectoralis muscles at the level of the nipple.

Scoring of sensation will be the following: 0= full sensation, 1= partial sensation, 2= no sensation (complete block) Following block placements, the subjects will be transported to the OR and general anesthesia will be induced. Following intubation, surgical procedure, emergence and extubation, the subject will be transported to the recovery room. In the recovery room or via phone post-discharge, at the 6 hour mark post-block placement, we will ask the subject if they are having any axillary pain. The severity of pain will be determined using the Numerical Rating Scale of 0-10. Zero is no pain and 10 is the most pain possible. Total opiate and benzodiazepine doses will be charted for the preoperative, intraoperative and PACU time frames.

ELIGIBILITY:
Inclusion Criteria:

* Adults, between 18 and 80 years of age
* Ability to take pills
* Agreement to a regional with general anesthesia technique

Exclusion Criteria:

* Allergy to amide local anesthetics
* Presence of a progressive neurological deficit
* pre-existing coagulopathy
* Current infection
* Significant pulmonary disease contraindicating phrenic nerve blockade
* Chronic use of an opioid analgesic (>3 months of a combined total of more than 40mg oxycodone equivalents a day)
* Inability to obtain ultrasound images of anatomy due to obesity.
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J.Wells Reynolds, MD, Principal Investigator — Wake Forest Baptist Health Department of Anesthesiology
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reynolds JW, Henshaw DS, Jaffe JD, Dobson SW, Edwards CJ, Turner JD, Weller RS, Graves BR, Freehill MT. Analgesic Benefit of Pectoral Nerve Block II Blockade for Open Subpectoral Biceps Tenodesis: A Randomized, Prospective, Double-Blinded, Controlled Trial. Anesth Analg. 2019 Aug;129(2):536-542. doi: 10.1213/ANE.0000000000004233. PMID 31136331

RESULTS

PARTICIPANT FLOW:
Groups:
- Interscalene Block Plus Sham Block: Twenty subjects will receive an ultrasound guided interscalene nerve block using the Solution for Injection in Interscalene Block dosed at the upper trunk location near the 6th cervical vertebral level, per standard clinical practice. A Sham Block of in area of PECS "Pectoralis" block will be done to allow for assessment of the intervention. Using the Solution for Injection in Sham Block.
  Interscalene Block: An interscalene block will be performed on the subjects.
  Sham Block
  Solution for Injection in Interscalene Block: 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine
  Solution for Injection in Sham Block: Lidocaine 1%
- Interscalene Plus PECS Blocks: Twenty patients will receive an ultrasound guided interscalene nerve block with Solution for Injection for Interscalene Block dosed at the 6th cervical root level, per standard clinical practice. Intervention subjects will also get a PECS "Pectoralis" 1 and 2 Blocks using the Solution for Injection PECS Blocks, dosed at the PECS1 location and PECS2 location as described by Blanco, et al.
  PECS "Pectoralis" 1 and 2 Blocks: An interscalene and a PECS "Pectoralis" 1 and 2 block will be performed on the subjects.
  Interscalene Block: An interscalene block will be performed on the subjects.
  Solution for Injection in Interscalene Block: 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine
  Solution for Injection PECS Blocks: 10mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at the PECS1 location and 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at PECS II.
Period: Overall Study
Arm/Group | Interscalene Block Plus Sham Block | Interscalene Plus PECS Blocks
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1
Not completed — Surgery type changed intra-operatively | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Interscalene Plus PECS Blocks: Twenty patients will receive an ultrasound guided interscalene nerve block using the Solution for Injection in Interscalene Block dosed at the upper trunk location near the 6th cervical vertebral level, per standard clinical practice. Intervention subjects will also a PECS "Pectoralis" II using the Solution for Injection PECS Blocks, dosed at the PECS1 location and PECS2 location as described by Blanco, et al.
  PECS "Pectoralis" II Blocks: An interscalene and a PECS "Pectoralis" 1 and 2 block will be performed on the subjects.
  Interscalene Block: An interscalene block will be performed on the subjects. Solution for Injection in Interscalene Block: 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine Solution for Injection PECS II Blocks: 10mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at the PECS1 location and 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at the PECS2 location.
- Total: Total of all reporting groups
Arm/Group | Interscalene Block Plus Sham Block | Interscalene Plus PECS Blocks | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 13 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 15 | 17 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Weight (kg) [Mean (Standard Deviation); unit: kg] | 88.1 (17.7) | 80.7 (18.2) | 84.3 (18.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (4.44) | 26.9 (4.55) | 27.8 (4.55)
Surgical Side (L/R) [Count of Participants; unit: Participants]
  Left sided surgery | 10 | 10 | 20
  Right sided surgery | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Axillary Pain
Description: Post-operative ambulatory surgery subjects will be asked 6 hours after block placement about the presence of axillary pain at rest. Numerical Rating Scale scores (0-10) will be recorded with 0= no pain, 10=most pain possible. Higher scores denotes worse outcome.
Time Frame: 6 hours post-block.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Interscalene Plus PECS Blocks: Twenty patients receive an ultrasound guided interscalene nerve block with Solution for Injection in Interscalene Block dosed at the upper trunk near the 6th cervical vertebral level, per standard clinical practice. For the Intervention, these subjects will also a PECS "Pectoralis" 1 and 2 Blocks using the Solution for Injection PECS Blocks, dosed at the PECS1 location and PECS2 location as described by Blanco, et al.
  PECS "Pectoralis" 1 and 2 Blocks: An interscalene and a PECS "Pectoralis" 1 and 2 block will be performed on the subjects.
  Interscalene Block: An interscalene block will be performed on the subjects.
  Solution for Injection in Interscalene Block: 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine
  Solution for Injection PECS Blocks: 10mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at the PECS1 location and 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at the PECS2
Arm/Group | Interscalene Block Plus Sham Block | Interscalene Plus PECS Blocks
Number analyzed (Participants) | 18 | 19
units on a scale | 3 [0 to 5.25] | 0 [0 to 1.5]

2. Secondary Outcome: Numerical Rating Scale Pain Scores (0-10) at Rest
Description: Subjects were asked about their overall shoulder pain during the followup phone call at 24hrs post-block. Numerical Rating Scale scores (0-10) will be recorded with 0= no pain, 10=most pain possible. Higher scores denotes worse outcome.
Time Frame: Assessed 24hrs post-block on a scale from 0-10.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Interscalene Block Plus Sham Block | Interscalene Plus PECS Blocks
Number analyzed (Participants) | 18 | 19
units on a scale | 6 [5 to 7] | 6 [4 to 7]

3. Secondary Outcome: Percentage of Participants With Episodes of Nausea or Vomiting
Description: Any episodes during the first 24 hours will be recorded as a yes.
Time Frame: Assessed 24hrs post-block (yes/no)
Measure: Number; unit: percentage of participants
Arm/Group | Interscalene Block Plus Sham Block | Interscalene Plus PECS Blocks
Number analyzed (Participants) | 18 | 19
percentage of participants | 39 | 37

4. Secondary Outcome: Total Opioid Usage
Description: Recorded in oxycodone equivalents in the first 24 hours post-discharge from the PACU.
Time Frame: Assessed 24hrs post-block in mg
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Interscalene Block Plus Sham Block | Interscalene Plus PECS Blocks
Number analyzed (Participants) | 18 | 19
mg | 31.6 [24.1 to 39.0] | 26.9 [21.8 to 32.0]

5. Secondary Outcome: Time From Block Placement to Onset of Axillary Pain
Description: Time self-reported by patients in the Interscalene Plus PECS Blocks group during data collection phone call at 24 hours post-block.
Time Frame: Assessed 24hrs post-block in hours
Population: This Outcome Measure was assessed only in the Interscalene Plus PECS Blocks group
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | Interscalene Plus PECS Blocks
Number analyzed (Participants) | 8
Hours | 16.7 [14.1 to 19.3]

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Interscalene Plus PECS Blocks: Twenty patients receive an ultrasound guided interscalene nerve block with Solution for Injection in Interscalene Block dosed at the upper trunk near the 6th cervical vertebral level, per standard clinical practice. For the Intervention, these subjects will also a PECS "Pectoralis" 1 and 2 Blocks using the Solution for Injection PECS Blocks, dosed at the PECS1 location and PECS2 location as described by Blanco, et al.
  PECS "Pectoralis" 1 and 2 Blocks: An interscalene and a PECS "Pectoralis" 1 and 2 block will be performed on the subjects.
  Interscalene Block: An interscalene block will be performed on the subjects.
  Solution for Injection in Interscalene Block: 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine
  Solution for Injection PECS Blocks: 10mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at the PECS1 location and 20mL of 0.25% bupivacaine with 1:400,000 epinephrine and 1:600,000 clonidine dosed at t
Arm/Group | Interscalene Block Plus Sham Block | Interscalene Plus PECS Blocks
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19

LIMITATIONS AND CAVEATS:
Only 8 patients in the PECS group reported the onset of axillary pain at home, so that data set is very limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT02741713/Prot_SAP_000.pdf